CLINICAL TRIAL: NCT06339424
Title: Investigation of Antitumor Immune Response in Patients With Unresectable Hepatocellular Carcinoma Undergoing Photon Radiotherapy Combined With Atezolizumab and Bevacizumab
Brief Title: Atezolizumab and Bevacizumab With Photon Radiotherapy for Unresectable Hepatocellular Carcinoma
Acronym: PhotonAB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202400156A3
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Photon Radiotherapy; HCC; PD-L1; VEGF; Atezolizumab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab and bevacizumab with photon radiotherapy (Experimental): Patients undergo Atezolizumab and Bevacizumab with photon radiotherapy.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Radiation: Photon radiotherapy

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be administered as an IV infusion on Day 1 of each cycle, with cycles occurring every 3 weeks. The initial dose will be delivered over 60 (± 15) minutes, and if well-tolerated, subsequent infusions may be given over 30 minutes. For patients who achieve a complete response (CR) within one year of treatment, atezolizumab should be continuously used for a year. For patients who experience a partial response (PR), atezolizumab should be continued until achieving CR or experiencing progressive disease (PD). Patients with stable disease should receive atezolizumab for 6 months. In the case of PD, atezolizumab should be discontinued at the time when PD is confirmed.
Drug: Bevacizumab — Bevacizumab 15 mg/kg will be administered as an IV infusion on Day 1 of each 3-week cycle. The initial dose will be delivered over 90 minutes (±15 minutes), and if well-tolerated, subsequent infusions may be given over 60 minutes. For patients who achieve a complete response (CR) within one year of treatment, bevacizumab should be continuously used for a year. In the case of patients experiencing a partial response (PR), bevacizumab should be continued until achieving CR or experiencing progressive disease (PD). Patients with stable disease should receive bevacizumab for 6 months. In the event of PD, bevacizumab should be discontinued when PD is confirmed. Temporary withholding or dose reduction of bevacizumab is permitted if patients experience adverse events such as bleeding episodes, severe hypertension, or proteinuria at the discretion of the treating physician.
Radiation: Photon radiotherapy — * 39.6-72.6 Gy in 22 fractions for tumors ≤1 cm from the hepatic hilum, bowel, and heart.
  * 30-66 Gy in 10 fractions for tumors >1 cm from the hepatic hilum, bowel, and heart.
  * 27.5-50 Gy in 5 fractions using stereotactic body radiation therapy (SBRT) techniques

SUMMARY:
Atezolizumab (anti-programmed death-ligand 1; anti-PD-L1) in conjunction with bevacizumab (anti-vascular endothelial growth factor; anti-VEGF) has become the established standard first-line systemic treatment for unresectable hepatocellular carcinoma (HCC). Despite an improved objective response rate (ORR) of 27%, the majority of patients face HCC progression and liver failure [Finn et al., N Engl J Med 2020]. Developing a new combined treatment strategy to overcome resistance to anti-PD-L1 and anti-VEGF is essential to improve patient outcomes.

Radiation treatment (RT) is highly efficacious in controlling localized solid tumors and has become an integral component of the treatment algorithm for unresectable HCC. Importantly, a recent retrospective cohort described that RT combined with atezolizumab plus bevacizumab was associated with favorable median overall survival of 16.1 months (Manzar et al, Cancers 2022). Our preclinical study (Hsieh et al., Science Immunology 2022) revealed that RT combined with PD-L1/PD-1 blockade induces immunogenic cell death and tumor antigen cross-presentation in antigen-presenting cells, thereby potentiating the systemic antitumor T cell responses in murine tumor models. However, whether the combinatorial therapy with RT, atezolizumab, and bevacizumab can trigger synergistic antitumor effects and systemic immune mobilization has not yet been validated in clinical trials for unresectable HCC.

Both atezolizumab/bevacizumab and X-ray RT are approved treatment methods for unresectable HCC by the U.S. and Taiwan Food and Drug Administration (FDA). The present phase II non-randomized trial aims to prospectively document the therapeutic efficacy, safety, and immunological responses in patients with unresectable HCC treated with atezolizumab/bevacizumab combined with conventional photon radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a diagnosis of HCC that is deemed unsuitable for surgical resection or transplant. Participants may have multiple lesions with a total maximal tumor dimension of < 20 cm, and no one lesion > 15 cm. Diagnosis should be confirmed by at least 1 criterion listed below:

   * Histologically or cytologically proven diagnosis of HCC.
   * Typical arterial enhancement and delayed washout on multiphasic CT or MRI.
2. Age ≥18 years at the time of signing the informed consent document.
3. ECOG performance status 0-1.
4. Barcelona Clinic Liver Cancer (BCLC) stages Intermediate (B) or Advanced (C).
5. Child-Pugh score 5-6 liver function within 28 days of study registration.
6. Documented virology status of hepatitis B virus (HBV), as confirmed by screening HBV serology test.
7. Documented virology status of hepatitis C virus (HCV), as confirmed by screening HCV serology test.
8. Ability to understand and the willingness to sign a written informed consent document
9. Adequate bone marrow, liver, and renal function within 4 weeks before study registration

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelet count ≥ 50,000/μL
   * Total bilirubin < 2.5 mg/dL
   * Serum albumin >2.8 g/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN)
   * Prothrombin time ≤ 6 seconds prolonged
   * Serum creatinine ≤ 1.5 mg/dL

Exclusion Criteria:

1. Prior invasive malignancy unless disease-free for a minimum of 2 years
2. Prior radiotherapy to the region of the liver that would result in overlap of radiation therapy fields
3. Prior selective internal radiotherapy/hepatic arterial yttrium therapy, at any time
4. Untreated active hepatitis B or hepatitis C
5. Moderate to severe or intractable ascites
6. Presence of distant metastases that cannot be encompassed by photon radiotherapy
7. Untreated or incompletely treated esophageal or gastric varices
8. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
   * Myocardial infarction within the last 6 months prior to study entry
   * Acute bacterial or fungal infection requiring intravenous antibiotics within 28 days prior to study entry
   * A bleeding episode within 6 months prior to study entry due to any cause.
   * Thrombolytic therapy within 28 days prior to study entry.
   * Known bleeding or clotting disorder.
   * Uncontrolled psychotic disorder
9. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
10. Prior solid organ transplantation.
11. Prior or active autoimmune disease (AID) including autoimmune hepatitis, inflammatory bowel disease, myasthenia gravis, systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, and multiple sclerosis.
12. Prior or active thrombotic or bleeding disorders, hemoptysis, cerebral vascular accident, significant cardiac disease (ischemic or congestive heart failure), or gastrointestinal perforation.
13. Inability to treat all sites of disease by photon radiotherapy (such as extrahepatic metastases or massive liver tumors whereby the liver constraints cannot be met for covering all sites of liver tumors.)
14. Known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 12 months
  PFS is defined as the time from signing the informed consent to the first occurrence of disease progression or death from any cause (whichever occurs first) according to RECIST1.1.

SECONDARY OUTCOMES:
Local control (LC) | 12 months
  LC is defined as the time from signing the informed consent to the first occurrence of disease progression in the irradiated field according to RECIST1.1.
Time to progression (TTP) | 12 months
  TTP is defined as the time from signing the informed consent to the first occurrence of disease progression according to RECIST1.1.
Overall Response Rate (ORR) | 12 months
  ORR is defined as a complete or partial response according to RECIST1.1.
Overall survival (OS) | 12 months
  OS is defined as the time from signing the informed consent to death from any cause.
Incidence and severity of adverse events | 12 months
  Adverse events will be graded using CTCAE v5

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data (IPD) with other researchers requires IRB review and approval. Presently, we do not have a plan to provide IPD to other researchers